CLINICAL TRIAL: NCT00340769
Title: Prevalence of a Non-Expressing 11B Mutation in Aka Peoples of the Central African Republic
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901160; 01-E-N160
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-12-20

CONDITIONS: Zinc Fingers Proteins
Keywords: Cytokines; Inflammation; mRNA Stability; Pygmy; Zinc Finger Proteins; Ethnic Group
MeSH Terms: conditions — Inflammation

SUMMARY:
The CCCH tandem zinc finger proteins are members of a small family of proteins that regulate the stability of certain types of mRNA containing so-called class II AU-rich elements in their 3'-untranslated regions. The best studied member of this protein family, tristetraprolin (TTP), exerts this destabilizing effect on at least two mRNAs coding for physiologically and medically important cytokines, tumor necrosis factor alpha and granulocyte macrophage colony stimulating factor. The physiological functions of the other two members of this protein family in mammals, 11B and 11D, are not known, but in experimental transfection studies they too can destabilize mRNAs containing this type of AU-rich element.

As part of the Environmental Genome Project, we resequenced the protein coding portions of the human genes encoding these three proteins, and uncovered a dinucleotide splice site mutation in the 11B gene in one of 144 alleles sequenced. We showed that this mutation created a novel restriction fragment length polymorphism, and that this mutation resulted in the failure of splicing and expression of the mRNA encoded by the mutant allele. Based on our previous data with mice completely deficient in TTP, we anticipate that complete deficiency of this protein, and possibly its partial deficiency, would result in human disease.

The mutant allele was from an anonymous adult Aka Pygmy women from the Central African Republic. We propose to genotype up to 1000 members of this ethnic group after obtaining buccal cell DNA from them. This will give us an approximate idea of the prevalence of this mutation in this population. If the mutation is found in a significant number of living individuals in this initial screen, then we will propose a later study of the individuals who have this genotype and their families. This second study, which will be reviewed separately, will attempt to correlate this genotype with a human trait or phenotype and possible y treatable human disease.

DETAILED DESCRIPTION:
The CCCH tandem zinc finger proteins are members of a small family of proteins that regulate the stability of certain types of mRNA containing so-called class II AU-rich elements in their 3'-untranslated regions. The best studied member of this protein family, tristetraprolin (TTP), exerts this destabilizing effect on at least two mRNAs coding for physiologically and medically important cytokines, tumor necrosis factor alpha and granulocyte macrophage colony stimulating factor. The physiological functions of the other two members of this protein family in mammals, 11B and 11D, are not known, but in experimental transfection studies they too can destabilize mRNAs containing this type of AU-rich element.

As part of the Environmental Genome Project, we resequenced the protein coding portions of the human genes encoding these three proteins, and uncovered a dinucleotide splice site mutation in the 11B gene in one of 144 alleles sequenced. We showed that this mutation created a novel restriction fragment length polymorphism, and that this mutation resulted in the failure of splicing and expression of the mRNA encoded by the mutant allele. Based on our previous data with mice completely deficient in TTP, we anticipate that complete deficiency of this protein, and possibly its partial deficiency, would result in human disease.

The mutant allele was from an anonymous adult Aka Pygmy women from the Central African Republic. We propose to genotype up to 1000 members of this ethnic group after obtaining buccal cell DNA from them. This will give us an approximate idea of the prevalence of this mutation in this population. If the mutation is found in a significant number of living individuals in this initial screen, then we will propose a later study of the individuals who have this genotype and their families. This second study, which will be reviewed separately, will attempt to correlate this genotype with a human trait or phenotype and possible treatable human disease.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Both genders are eligible.

Ages included children through adulthood.

Must be willing and able to participate and understand the explanations and instructions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 2001-04-18; Study Completion 2006-12-20

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina
  - Washington State University, Vancouver, Washington
- Ministry of Health and Scientific Research, Bangui, Central African Republic